CLINICAL TRIAL: NCT06447493
Title: Exploring the Effects of Spencer's Technique on Shoulder Function: A Pilot Study
Brief Title: Effects of Spencer's Technique on Shoulder Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Daniel Cawley, Assistant Professor, Edward Via Virginia College of Osteopathic Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-061
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Shoulder
Keywords: Osteopathic Physicians; Shoulder; Diagnostic Imaging; Motion Capture; Range of Motion, Articular; Blood Circulation; Pain
MeSH Terms: conditions — Pain | interventions — RE1-silencing transcription factor

STUDY DESIGN:
Intervention Model Description: Two by Two cross-over trial. Measurements will be taken on both shoulders with only the dominant shoulder receiving osteopathic manipulative treatment (OMT). The order in which the measurements and OMT treatment is performed will be randomized. The cross-over design allows for the opportunity to estimate 3 components, the possible effect of ultrasound measurement on the outcomes even when OMT is not performed, the combined effect of OMT and ultrasound measurements on outcomes, and an adjusted estimate OMT treatment effect removing any ultrasound effects if those effects exist. Change scores for all outcomes will be calculated per shoulder and then a comparison between change scores will be conducted using a paired design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OMT Intervention, then Rest (Experimental): 10 subjects will be randomized to begin with the dominant shoulder. Investigators will measure baseline outcomes on the dominant shoulder, apply OMT treatment, measure post treatment outcomes on dominant shoulder, a 5-minute rest period as a washout period, then proceed to measure baseline measures on non-dominant shoulder, a rest that is equivalent to the time needed for OMT treatment, ending with post measurements on the non-dominant shoulder.
  Interventions: Other: Osteopathic Manipulative Treatment-Spencer's Technique (Modified); Other: Rest
- Rest, then OMT Intervention (Experimental): 10 subjects will be randomized to begin with the non-dominant shoulder. Investigators will measure baseline outcomes on the non-dominant shoulder, a rest period equivalent to the time needed for OMT treatment, measure post treatment outcomes on non-dominant shoulder, a 5-minute rest period as a washout period, then proceed to measure baseline measures on dominant shoulder, provide OMT treatment, ending with post measurements on the dominant shoulder.
  Interventions: Other: Osteopathic Manipulative Treatment-Spencer's Technique (Modified); Other: Rest

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment-Spencer's Technique (Modified) — Combination OMT approach utilizing Muscle Energy Technique (MET), Articulatory Technique (ART), and Myofascial Release (MFR). It is a series of direct OMT addressing the barrier of somatic dysfunction (SD) with the goal of restoring neurovascular balance and improved motion of the shoulder girdle and glenohumeral joint. Utilizing these three OMT techniques, the practitioner attempts restoration of glenohumeral joint motion using shoulder extension, flexion, circumduction with compression, circumduction with distraction, abduction, adduction, external rotation, internal rotation, and distraction in abduction. The study uses a modified version of the Spencer technique, done in the seated position for patient comfort, as well as adding to the treatment sequence: latissimus dorsi, pectoralis minor-major, serratus anterior, and rhomboid major-minor. Adding these muscles into treatment will help to address and correct sternoclavicular joint SD, acromioclavicular joint SD, and scapular SD.
Other: Rest — 10 minute rest period.

SUMMARY:
The purpose of this study is to see the impact of a modified Spencer's technique on tissue stiffness, mobility, and blood flow of the shoulder joint. Spencer's technique is a well-known osteopathic manipulative treatment (OMT) that is common for treating adhesive capsulitis and is believed to help blood flow. There are studies that look at the clinical effects of the technique and/or compare it to other techniques; however, measuring the extent to which Spencer's technique, or this modified technique, improves tissue stiffness and blood flow has never been written in the literature. This study will serve as a proof of concept that this technique improves tissue stiffness, blood flow, and mobility of the shoulder join as well as the nearby areas. Using ultrasound, the investigators will measure tissue stiffness and blood flow and will analyze the mobility of the shoulder joint using a Vicon motion capture system.

ELIGIBILITY:
Inclusion Criteria:

• male and female subjects 18-50 years old

Exclusion Criteria:

* prior shoulder surgery or injury to the reported dominant throwing arm
* shoulder pain in the reported dominant throwing arm within the last 6 months
* diagnosis cervical radiculopathy or pinched nerve in the neck
* connective tissue or muscle disorders
* known pregnancy
* tobacco use
* known diabetes or prediabetes
* allergy to ultrasound gel (propylene glycol)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Muscle Stiffness | Day 1 Pre, Day 1 Post, Day 2
  Using Shear Wave Elastography to measure muscle stiffness (kPa) of the supraspinatus, infraspinatus, posterior shoulder capsule, and coracoacromial ligament.
Shoulder Mobility | Day 1 Pre, Day 1 Post, Day 2
  Using Vicon motion capture system to calculate landmark coordinates and using morphometric canonical variate analysis to analyze mobility changes.
Microvascular/capillary blood flow | Day 1 Pre, Day 1 Post, Day 2
  Using ultrasound to capture blood flow of the supraspinatus, infraspinatus, posterior shoulder capsule, and coracoacromial ligament.
Subjective Shoulder Stiffness (Visual Analogue Scale) | Day 1 Pre, Day 2
  Using Visual Analogue scale to measure participant's subjective measure of shoulder stiffness. Scores range from 0 to 10, with 0 being "Not stiff at all" and 10 being "Very stiff."

CONTACTS AND LOCATIONS:
Locations (1):
- Edward Via College of Osteopathic Medicine-Auburn, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knebl JA, Shores JH, Gamber RG, Gray WT, Herron KM. Improving functional ability in the elderly via the Spencer technique, an osteopathic manipulative treatment: a randomized, controlled trial. J Am Osteopath Assoc. 2002 Jul;102(7):387-96. PMID 12138953
- [Background] Iqbal M, Riaz H, Ghous M, Masood K. Comparison of Spencer muscle energy technique and Passive stretching in adhesive capsulitis: A single blind randomized control trial. J Pak Med Assoc. 2020 Dec;70(12(A)):2113-2118. doi: 10.5455/JPMA.23971. PMID 33475581
- [Background] Haveela, B., Praveen Dowle, and P. Chandrasekhar.
- [Background] Yamaguchi K, Sher JS, Andersen WK, Garretson R, Uribe JW, Hechtman K, Neviaser RJ. Glenohumeral motion in patients with rotator cuff tears: a comparison of asymptomatic and symptomatic shoulders. J Shoulder Elbow Surg. 2000 Jan-Feb;9(1):6-11. doi: 10.1016/s1058-2746(00)90002-8. PMID 10717855
- [Background] Kunz P, Mick P, Gross S, Schmidmaier G, Zeifang F, Weber MA, Fischer C. Contrast-Enhanced Ultrasound (CEUS) as Predictor for Early Retear and Functional Outcome After Supraspinatus Tendon Repair. J Orthop Res. 2020 May;38(5):1150-1158. doi: 10.1002/jor.24535. Epub 2019 Dec 2. PMID 31769543
- [Background] Matava MJ, Purcell DB, Rudzki JR. Partial-thickness rotator cuff tears. Am J Sports Med. 2005 Sep;33(9):1405-17. doi: 10.1177/0363546505280213. PMID 16127127
- [Background] Lawrence RL, Moutzouros V, Bey MJ. Asymptomatic Rotator Cuff Tears. JBJS Rev. 2019 Jun;7(6):e9. doi: 10.2106/JBJS.RVW.18.00149. PMID 31246863
- [Background] Coren S. Measurement of handedness via self-report: the relationship between brief and extended inventories. Percept Mot Skills. 1993 Jun;76(3 Pt 1):1035-42. doi: 10.2466/pms.1993.76.3.1035. PMID 8321574